CLINICAL TRIAL: NCT01085656
Title: A Phase I Clinical Trial of OXi4503 for Relapsed and Refractory Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndromes (MDS)
Brief Title: A Phase I Clinical Trial of OXi4503 for Relapsed and Refractory AML and MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF OXi4503 AML MDS
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Leukemia, Myelogenous, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Oxi 4503

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OXi4503 (Experimental): Dosing of OXi4503 will be an intravenous infusion (IV) over 10 minutes on Days 1, 8, 15, and 22 of each 28 day cycle.
  Interventions: Drug: OXi4503

INTERVENTIONS:
Drug: OXi4503 — Two safety cohorts treating two (2) patients at a dose of 2.5 mg/m2 followed by two patients at 3.75 mg/m2 will be completed prior to beginning at the dose level of 5 mg/m2.
  Dosing of OXi4503 will be an intravenous infusion (IV) over 10 minutes on Days 1, 8, 15, and 22 of each 28 day cycle.
  Dose escalations and de-escalations of 25% will be made until the maximum tolerated dose is reached.
  Number of cycles: After Cycle 1, subjects who achieve stable disease (SD) or greater response may continue to receive additional cycles of treatment until either disease progression (defined as greater than 25% increase in leukemia myeloblasts in the bone marrow compared to baseline examination) or unacceptable toxicity due to the investigational agent.
  Other Names: Combretastatin A1 Diphosphate, CA1P

SUMMARY:
This study is intended to determine the safety and maximum tolerated dose of a drug, OXi4503 (combretastatin A1 diphosphate, CA1P, OXiGENE), in patients with relapsed and refractory AML and MDS.

DETAILED DESCRIPTION:
Despite initial disease remissions with cytotoxic chemotherapies, patients with AML and MDS often relapse and die of their disease. Novel strategies for targeting dependent pathways are needed. AML and MDS depend on blood vessels for survival and proliferation. OXi4503 is a novel microtubule targeting agent that selectively destroys cancer-associated blood vessels, induces cancer cell apoptosis via an ortho-quinone moiety and results in significant regressions of solid tumors. OXi4503 is currently being tested in phase I clinical trials of advanced solid tumors. In preclinical studies with human AML, OXi4503 was cytotoxic to leukemia cells, decreased size of chloromas, regressed leukemic cell engraftment in bone marrow and brought about phenotypic and molecular remissions. Given these results, we hypothesize that OXi4503 has disease remitting effects in myeloid malignancies such as AML and MDS. Before evaluating efficacy, safety and maximum tolerated dose of OXi4503 will be defined in AML and MDS patients. In addition, assessments of pharmacokinetic (PK) and pharmacokinetic (PD) parameters will be made, and relationships between dose and biologic activity will be defined. Results from this trial will provide new clinical data and biologic insight regarding the effects of OXi4503 in AML and MDS, and will serve as the basis for future efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age;
* Patients must have either:

  * AML (de novo or secondary, and any WHO 2008 classification excluding acute promyelocytic leukemia) that has failed to achieve CR or CRi (IWG 2003) after at least 1 cycle of induction chemotherapy, or has relapsed after any duration of CR or CRi; or,
  * MDS (RAEB-1 or RAEB-2 WHO 2008 classification) that has failed to achieve any hematologic improvement (IWG 2006 criteria) after at least 4 cycles of induction therapy (e.g., azacitidine, decitabine), or has relapsed after any duration of CR or PR.;
* Patient performance status must be Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2;
* Patients must have a life expectancy of greater than 14 days;
* Patients must have total bilirubin ≤ 2;
* Patients must have serum AST and ALT levels ≤ 2.5 times upper limit of normal;
* Patients must have serum creatinine less than or equal to 2.5 times upper limit of normal;
* Patients must have PT/INR and PTT in normal range ± 25%;
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) may participate, provided they meet the following conditions:

  * Must agree to use physician-approved contraceptive methods (e.g., abstinence, intrauterine device, oral contraceptive, double barrier device) throughout the study and for three months following the last dose of OXi4503; and
  * Must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial;
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 6 months following the last dose of OXi4503;
* Written informed consent, willingness, and ability to comply with all study procedures.

Exclusion Criteria:

* Acute promyelocytic leukemia (APL) with t(15;17);
* Absolute peripheral blood myeloblast count greater than 25,000/mm3;
* Uncontrolled hypertension, defined as blood pressure 140/90 mm Hg despite maximum medical intervention;
* History of congenital long QT syndrome or torsades de pointes;
* Pathologic bradycardia or heart block (excluding first degree heart block);
* Prolonged baseline QTc, defined as QTc interval > 470 msec in women and > 450 msec in men;
* History of ventricular arrhythmia (excluding premature ventricular contractions, PVCs);
* Major operative surgery within 28 days;
* Unstable angina pectoris within 28 days;
* Myocardial infarction and/or new ST elevation or depression or new Q wave on ECG within 28 days;
* Any history of hemorrhagic stroke;
* Symptomatic congestive heart failure Class III or greater (New York Heart Association Functional Classification);
* On full dose anti-coagulation defined as warfarin intended to raise the INR to 2-3, or enoxaparin 1 mg/kg twice a day or unfractionated heparin intended to raise the PTT to 60-90 seconds;
* Major hemorrhagic event within 28 days requiring transfusion of packed red blood cells;
* Prior history of hypertensive crisis or hypertensive encephalopathy;
* Active, uncontrolled, clinical significant infection;
* Any open wound;
* Pregnant and nursing patients are excluded because the effects of OXi4503 on a fetus or nursing child are unknown.
* Treatment with any anticancer therapy (standard or investigational) within the previous 21 days prior to the first dose of study drug or less than full recovery (CTCAE grade 1) from the clinically significant toxic effects of that treatment. The use of hydroxyurea may be used for two weeks after dosing in Cycle 1 (e.g., Days 1-14 dosed with hydroxyurea).

Relative Exclusion Criteria:

* Patients on concurrent medications known to prolong the QTc interval may participate as long as their screening QTc interval meets eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and establish the maximum tolerated dose (MTD) of OXi4503 in patients with relapsed and refractory AML and MDS. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Cogle, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Cancer Hopsital, Gainesville, Florida, United States